CLINICAL TRIAL: NCT06966544
Title: Investigating the Effectiveness of Graded Motor Imagery Training on Upper Limb Function, Proprioception, Functional Mobility, Balance and Quality of Life in Children With Obstetric Brachial Plexus Injury
Brief Title: Investigating the Effectiveness of Graded Motor Imagery Training in Children With Obstetric Brachial Plexus Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Hüseyin MAHİROĞLU, PhD Student, Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BakircayU-FTR-HM-01
Record Dates: First submitted 2025-05-04; First posted 2025-05-12 (Actual); Last update posted 2025-05-12 (Actual); Status verified 2025-05

CONDITIONS: Obstetric Brachial Plexus Injury

STUDY DESIGN:
Intervention Model Description: Two groups; conventional physiotherapy versus conventional physiotherapy plus graded motor imagery training.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Physiotherapy Group (Active Comparator): Participants were randomly divided into two arms. Participants in the activate comparator group will be administered traditional physiotherapy approaches applied after obstetric brachial plexus injury by the researcher physiotherapist.
  Interventions: Other: Conventional Physiotherapy
- Graded Motor Imagery Group (Experimental): Participants included in the motor imagery group through randomization will receive a progressive motor imagery approach in addition to the conventional physiotherapy treatment received by the first group. All applications are performed by the same physiotherapist.
  Interventions: Other: Graded Motor Imagery

INTERVENTIONS:
Other: Conventional Physiotherapy — All subjects to be included in our study were evaluated before and after treatment by a physiotherapist acting as a blinded evaluator. In the treatment, conventional physiotherapy approaches are applied twice a week for 8 weeks by the physiotherapist conducting the thesis study. In parallel with the initial evaluation, an individualized conventional physiotherapy program is created according to the functional status of the children and the severity and type of the affected area.
  The main topics of this program consist of the following: Normal range of motion exercises for shoulder, elbow, wrist and fingers, strengthening exercises for scapulothoracic, shoulder, elbow, hand-wrist joints in all directions, stretching exercises for shoulder, elbow, wrist, fingers (to be selected depending on the patient's involvement), scapulothoracic mobilization, glenohumeral mobilization and elbow according to possible limitations, hand-wrist joint mobilization techniques (myofascial release, gliding
  Arms: Conventional Physiotherapy Group
Other: Graded Motor Imagery — All approaches applied to the conventional physiotherapy group are applied to this group in the same manner and duration (8 weeks-twice a week). However, in addition to conventional physiotherapy, progressive motor imagery (AMI) training program is being applied twice a week for 8 weeks.
  In the GMI program, in addition to this program, components of GMI training will be applied to sequentially activate cortical motor networks and improve cortical organization. These are;
  * Laterality training with the help of visuals selected in the first stage (0-2 weeks)
  * In the second stage, motor imagery activities designed in the form of scenarios to be developed specifically for motor activity deficiencies seen in OBPY (2-5 weeks)
  * In the third stage, a mirror therapy program will be prepared (5-8 weeks).
  Arms: Graded Motor Imagery Group

SUMMARY:
The aim of this study is to investigate the effect of graded motor imagery training on upper extremity motor function, proprioception, functional mobility, balance and quality of life in patients with obstetric brachial plexus injury in addition to conventional treatment. In this context, our aim is to identify new and potential physiotherapeutic approaches to address deficits in motor planning that have been shown to occur at the level of the central nervous system.

DETAILED DESCRIPTION:
This study was planned as a randomized, controlled, single-blind study. The aim of this study was to investigate the effects of graded motor imagery (GMI) training, performed in addition to conventional treatment of patients with obstetric brachial plexus injury, on upper extremity motor function, proprioception, functional mobility and quality of life. In parallel to the initial assessment, a conventional physiotherapy program was created that is individualized according to the functional status and severity of the effects in the children. In the GMI program, in addition to this program, the components of GMI training are applied to sequentially activate the cortical motor networks and develop cortical organization. All assessments of the participants before and at the end of the treatment are carried out by a blind physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* Obtaining family consent and the child's willingness
* Being between the ages of 7-18
* Being diagnosed with obstetric brachial plexus injury
* Not having received physical therapy in the last 6 months

Exclusion Criteria:

* Having a traumatic (postnatal) brachial plexus injury
* Having undergone surgery for complications related to brachial plexus injury within the last six months (release, tendon transfer, osteotomy, etc.)
* Having another neurological, neuromuscular, musculoskeletal or cardiopulmonary system disease in addition to OBPI

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
The Modified Mallet Classification System | 8 weeks
  The modified Mallet classification is one of the valid and reliable scales frequently used in the literature to determine the functional status of the extremity in cases with brachial plexus lesions. This classification system aims to evaluate the global characteristics of the extremity rather than evaluating the functions of individual muscles. In this system, the extremity's global abduction, global external rotation, and the adequacy of the hand reaching the neck, mouth and back to the spine are evaluated. A score between 0 and 5 is made according to the position and degree of strain during each movement. The maximum score that can be obtained is 25, and the score obtained gives an idea about the functional status of the extremity.
Active Movement Scale | 8 weeks
  Prepared by the Brachial Plexus Clinic of The Hospital for Sick Children (Toronto). In the OBPY group, the affected upper extremity was evaluated with 15 joint movements (from the shoulder to the fingers) specified on the scale. The movement is first examined in the position where gravity is eliminated, and if a full score is obtained, it is evaluated in the position against gravity and a score between (0-7) is given.
The Quality of Upper Extremity Skills Test (QUEST) | 8 Weeks
  QUEST is a test that evaluates the child's manual skills and the quality of movement. It was developed by Prof. Dr. Carol De MATTEO for use in the 18-month-8 age group. Later, the validity and reliability study of this test was conducted for 4-12 age groups. There are studies in the literature regarding its use in children between the ages of 2-15. The sections of QUEST are as follows: A. Independent movements B. Grasping C. Weight bearing D. Protective extension E. Hand function rate F. Cooperation rates.
Range of Motion Measurement | 8 Weeks
  Range of motion will be assessed by measuring the range of motion of the shoulder, elbow and wrist joints with a universal goniometer. Active joint movements of the patients will be measured with a universal goniometer before and after treatment and recorded as degrees.

SECONDARY OUTCOMES:
Box and Block Test | 8 Weeks
  The Box and Block Test is a test developed to measure gross manual dexterity. It is a good indicator of the severity of upper extremity involvement in OBPY. In the study, the number of blocks collected in 60 seconds is calculated as in the original procedure of the test.
Proprioception Assessment | 8 Weeks
  For proprioceptive sense evaluation, joint position sense evaluation (angle reconstruction test) is used in shoulder and elbow joints. The joint to be measured is ensured to be seen clearly. Digital inclinometer is used to evaluate poprioceptive sense. Shoulder joint proprioceptive sense is performed three times at 60, 90 and 120 degree angles using active reposition test. Eyes are covered with a tape. It is brought from 0 degree starting position to target angles of and waited for 5 seconds for the individual to learn this position and placed back to the starting position. The individual is then asked to actively bring his arm to the previously taught target angle and this test is repeated 3 times for each target angle. After the test, the average of the three angles is taken for each target angle. Elbow joint flexion is evaluated as specified at 30, 60, 90° angles.
Timed Up and Go Test | 8 Weeks
  The Timed Up and Go Test is a simple, practical and rapid test used to assess functional mobility and dynamic balance. Children are asked to get up from a standard chair with back and arm support, walk a predetermined distance of 3 meters as fast as possible without running, return without touching anything, walk back to the chair and return to a sitting position. The time taken is recorded in seconds (sec).
Timed Stair Climb Test | 8 Weeks
  The Timed Stair Climbing and Descending Test is another test that has been proven to be valid and reliable in the assessment of functional mobility and dynamic balance. The test begins with the child standing 30 cm away from the bottom rung of a 10-step staircase and climbing the steps with the command. The individual is asked to climb the steps safely but as quickly as possible and then turn and descend without waiting after climbing the last step, and the test is completed when the individual descends the last step with both feet touching the ground. The test score is recorded as time (sec).
Functional Reach Test | 8 Weeks
  This test was developed to assess stability. The functional reach test is an easily applicable, performance-based assessment method. It is defined as the maximum distance that an individual can reach forward in the horizontal plane while maintaining stability on the support surface in a standing position. The person holds the shoulder parallel to the surface being measured while in 90-degree flexion. The distance between the shoulder and the tip of the 3rd finger is measured. Then, patients are asked to reach the farthest distance possible without moving their feet, and the point where the tip of the 3rd finger reaches is marked on the surface.
Quality of Life Assesment | 8 Weeks
  The pediatric quality of life scale (PedsQL 4.0) will be used to assess health-related quality of life. The scale was developed to assess the health-related quality of life of children and adolescents aged 2-18 and consists of 5 main headings. These are; physical functioning (8 items), emotional functioning (5 items), social functioning (5 items), and school functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Gulbin Ergin, Associate Professor, Study Director — İzmir Bakırcay University
Locations (1):
- Izmir Bakircay University Physiotherapy and Rehabilitation Application and Research Center, Izmir, Menemen, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
After the data collection, another study is planned in the future, which includes long-term follow-up related to the data.